CLINICAL TRIAL: NCT00288249
Title: Prospective, Multicenter, Randomized, Independent-group, Open-label Phase II Study to Investigate the Efficacy, Safety and Tolerability of 4 Regimen With 3 Doses of ZK 219477 (16 and 12 mg/m2 Body Surface Area as 3-hour Infusion or 22 mg/m2 Body Surface Area as 30-minute or 3-hour Infusion) in Patients With Metastatic Breast Cancer
Brief Title: Safety and Efficacy Study of a New Chemotherapy Agent to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91464; 2005-003216-30 (EudraCT Number); 309544 (Other: Company Internal)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Breast Neoplasms; Breast Cancer, Metastatic
Keywords: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 2 (Experimental): Each subject was scheduled to receive one infusion of ZK 219477 every 3 weeks in one of the respective arms (16 mg/m2 in Arm 1, 12 mg/m2 in Arm 2, 22 mg/m2 [30-minute infusion] in Arm 3 and 22 mg/m2 [3-hour infusion] in Arm 4)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)
- Arm 3 (Experimental): Each subject was scheduled to receive one infusion of ZK 219477 every 3 weeks in one of the respective arms (16 mg/m2 in Arm 1, 12 mg/m2 in Arm 2, 22 mg/m2 [30-minute infusion] in Arm 3 and 22 mg/m2 [3-hour infusion] in Arm 4)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)
- Arm 4 (Experimental): Each subject was scheduled to receive one infusion of ZK 219477 every 3 weeks in one of the respective arms (16 mg/m2 in Arm 1, 12 mg/m2 in Arm 2, 22 mg/m2 [30-minute infusion] in Arm 3 and 22 mg/m2 [3-hour infusion] in Arm 4)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)
- Arm 1 (Experimental): Each subject was scheduled to receive one infusion of ZK 219477 every 3 weeks in one of the respective arms (16 mg/m2 in Arm 1, 12 mg/m2 in Arm 2, 22 mg/m2 [30-minute infusion] in Arm 3 and 22 mg/m2 [3-hour infusion] in Arm 4)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)

INTERVENTIONS:
Drug: Sagopilone (BAY86-5302, ZK 219477) — 16 mg/m2, 3-hour i.v. infusion, 1 cycle every 3 weeks. Planned number of cycles : 2-6.
  Arms: Arm 1
Drug: Sagopilone (BAY86-5302, ZK 219477) — 12 mg/m2, 3-hour i.v. infusion, 1 cycle every 3 weeks. Planned number of cycles : 2-6.
  Arms: Arm 2
Drug: Sagopilone (BAY86-5302, ZK 219477) — 22 mg/m2, 30-minute i.v. infusion, 1 cycle every 3 weeks. Planned number of cycles : 2-6.
  Arms: Arm 3
Drug: Sagopilone (BAY86-5302, ZK 219477) — 22 mg/m2, 3-hour i.v. infusion, 1 cycle every 3 weeks. Planned number of cycles : 2-6.
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine whether the study drug is effective and safe in the treatment of patients with metastatic breast cancer

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer
* No previous treatment with taxanes, and vinca alkaloids
* Use of highly effective birth control methods in females of child-bearing potential

Exclusion Criteria:

* More than 2 previous chemotherapies
* Previous participation in another trial within the last 4 weeks
* Breast feeding
* Active infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-12; Primary Completion 2008-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (complete or partial response according to RECIST) | Every 6 weeks
  The proportion of subjects with either complete or partial response according to the modified RECIST criteria was calculated as best overall response after 6 courses of therapy (i.e., before Course 7).

SECONDARY OUTCOMES:
Duration of complete or partial tumor response | Every 6 weeks
  Defined as the time between the first date that confirmed complete or partial response was established as "overall response" and the first date that recurrence or overall response of progressive disease was documented
Time to tumor progression | Every 6 weeks
  Defined as the time from the start of study treatment to the first objective evidence of tumor progression, symptomatic deterioration, or death from cancer

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Vienna, Vienna, Austria
- Brasschaat, Belgium
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- France (5):
  - Vandœuvre-lès-Nancy, France
  - Angers
  - Bordeaux
  - Clermont-Ferrand
  - Saint-Herblain
- Berlin, State of Berlin, Germany
- Italy (3):
  - Forlì, FC
  - Milan, MI
  - Reggio Emilia, RE
- Poland (2):
  - Olsztyn
  - Warsaw
- Ljubljana, Slovenia
- Spain (2):
  - Madrid, Madrid
  - Málaga, Málaga
- Manchester, Greater Manchester, United Kingdom